CLINICAL TRIAL: NCT00185419
Title: An Open-Label, Randomised, Parallel-Group Comparison to Investigate the Efficacy of Yasmin® (30 µg Ethinylestradiol, 3mg Drospirenone) and Marvelon® (30 µg Ethinylestradiol, 150 µg Desogestrel) on Cycle Control in Healthy Chinese Women Over 13 Cycles
Brief Title: A Clinical Study on Yasmin® vs. Marvelon® in Chinese Women Requiring Contraception
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 91330; 308062
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Contraception
MeSH Terms: interventions — drospirenone and ethinyl estradiol combination; Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Yasmin
- Arm 2 (Active Comparator)
  Interventions: Drug: Marvelon

INTERVENTIONS:
Drug: Yasmin — 30 µg ethinylestradiol, 3mg drospirenone
  Arms: Arm 1
Drug: Marvelon — 30 µg ethinylestradiol, 150 µg desogestrel
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness in terms of prevention of pregnancy and safety of the oral contraceptive Yasmin and Marvelon on cycle control in healthy Chinese women

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese female requesting contraceptives

Exclusion Criteria:

* Vascular, metabolic, hepatic, renal, oncologic and other diseases

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 842 (Actual)
Dates: Start 2003-11; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the comparison of cycle control from randomisation to cycle 13. This will be based on the number of subjects reporting at least 1 unexpected intracyclic bleeding episode between cycles 2 to 13. | 13 treatment cycles (1 cycle= 28 days)

SECONDARY OUTCOMES:
Weight changes | 13 treatment cycles
Contraceptive reliability | 13 treatment cycles
Effects on skin condition | 13 treatment cycles
Changes in MDQ subscale scores | 13 treatment cycles
Adverse Events | the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Ask Contact, China